CLINICAL TRIAL: NCT05261100
Title: Effects of Routine Physical Therapy With and Without Core Stability Exercises in Patients With Patellofemoral Pain Syndrome -a Randomized Controlled Trial
Brief Title: Effects of Core Stability Exercises in Patients With Patellofemoral Pain Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lahore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: ULahore Hassan javed
Record Dates: First submitted 2022-02-19; First posted 2022-03-02 (Actual); Last update posted 2022-06-28 (Actual); Status verified 2022-06

CONDITIONS: Patellofemoral Pain Syndrome
Keywords: Patellofemoral Pain Syndrome; Core stability
MeSH Terms: conditions — Patellofemoral Pain Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active group (Placebo Comparator): Conventional Physical therapy
  Interventions: Other: Conventional Physical Therapy
- Experimental group (Experimental): Conventional Physical therapy with Core stability
  Interventions: Other: Core stability exercises

INTERVENTIONS:
Other: Core stability exercises — Moist heating pads will be applied on knee joint for 10 minutes before each treatment session.
  Apply TENS on knee joint for 10 minutes treatment session. Knee Isometric exercises will be performed along with core stability exercises..
  Other Names: Conventional Physical Therapy
  Arms: Experimental group
Other: Conventional Physical Therapy — Moist heating pads will be applied on knee joint for 10 minutes before each treatment session.
  Apply TENS on knee joint for 10 minutes treatment session. Knee Isometric exercise perform.
  Arms: Active group

SUMMARY:
The purpose of the study is to compare the effects of routine physical therapy with and without core stability exercises on pain and range of motion, in patients with patellofemoral pain syndrome. The spine, abdominal region, pelvis, hips, and proximal lower extremities, are defined as the core of the body. The effects of core muscle strengthening have been proven as an effective method of management in various cases. The knee is the frequently injured joint in core instability with the decreased hip strength. Deficiency in the control of the neuromuscular system of the body's trunk or "core" may affect the stability of the lower extremity, which can lead to injury in the tibiofemoral or patellofemoral joints.

DETAILED DESCRIPTION:
The patellofemoral pain syndrome (PFPS) is a common cause for "anterior knee pain" and mainly affects young women without any structural changes such as increased Q-angle or significant pathological changes in articular cartilage. Patellofemoral pain syndrome (PFPS) is the most common overuse syndrome in athletes. Patellofemoral pain is more common among female athletes especially adolescents and young adults. Symptoms include: persistent pain behind the patella or peripatellar. Pain increases on ascending and descending stairs and squatting and prolonged sitting.

Patellofemoral Pain Syndrome (PFPS) is a common musculoskeletal disorder typically occurring in physically active people aged 40 years and younger, causing pain, functional deficits and lower limb weakness. Traditional treatment has been aimed at strengthening the knee, however recent research suggests the muscles around the hip also play an important role in the development and continuity of Patellofemoral Pain Syndrome.

Patellofemoral pain (PFP) is pain in the peripatellar/retropatellar region that aggravates with physical activities such as squatting, stair climbing, running and jumping or sitting for prolonged periods of time. It is the most common source of anterior knee ailment in active adolescents and young adults and is much more prevalent in women than men.

Patellofemoral pain (PFP) is a very common problem in athletes who participate in jumping sports. Several risk factors may play a part in the pathogenesis of PFP. Overuse, trauma and intrinsic risk factors are particularly important among athletes. Physical examination has a key role in PFP diagnosis. common risk factors should be investigated, such as hip muscle dysfunction, poor core muscle endurance, muscular tightness, excessive foot pronation and patellar malalignment.

Studies conducted on core muscle strengthening exercises program for the management of pain in hip, quadriceps region and ankle joint but limited studies were conducted in patient with patellofemoral pain syndrome. There is a need to compare the effectiveness of routine physiotherapy with and without core stability exercises in patient with patellofemoral pain syndrome. This study is intended to determine the effectiveness of core muscle strengthening exercises for the management of patellofemoral pain syndrome.

The spine, abdominal region, pelvis, hips, and proximal lower extremities, are defined as the core of the body. The effects of core muscle strengthening have been proven as an effective method of management in various cases. The knee is the frequently injured joint in core instability with the decreased hip strength. Deficiency in the control of the neuromuscular system of the body's trunk or "core" may affect the stability of the lower extremity, which can lead to injury in the tibiofemoral or patellofemoral joints.

ELIGIBILITY:
Inclusion Criteria:

* • Age between 18-40 Years

  * Both Gender
  * Patient with Anterior knee pain for at least 4 weeks

Exclusion Criteria:

* • History of trauma ,fracture of spine and lower extremity

  * History of any congenital deformity
  * History of lumbar radiculopathy
  * History of hip osteoarthritis
  * History of rheumatoid arthritis
  * History of Any surgical procedure involving lumber or lower extremity

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2021-11-11 (Actual); Primary Completion 2022-03-15 (Actual); Study Completion 2022-05-08 (Actual)

PRIMARY OUTCOMES:
Pain (Visual Analogue Scale) | 6 weeks
  The visual analogue scale is a simple and commonly used way for the assessment of variations in intensity of pain. In clinical practice the ratio of pain relief, evaluated by VAS, is frequently considered as a measure of the efficacy of treatment. VAS range is 0-10. It's a categorical scale with 0-4 mild pain, 4-7 moderate or distressing pain while 7-10 unbearable pain30. In this study inclusion criteria will be categorically 0-7 score, mild & moderate pain intensity on VAS. Use is scale for intensity of pain.
  Total eight treatment sessions will be given to each patient, and pre-treatment assessment will be done on very first day. Second assessment will be done on fourth treatment session, and final assessment will be on eighth treatment session.
Range of Motion (Goniometer) | 6 weeks
  A goniometer is a device used in physical therapy to measure a joint's range of motion (ROM). There are two "arms"-one that is stationary and one that is movable-that are hinged together.
  In order to assess the range of knee joint, goniometer will be used. Stationary arm will be placed on lateral epicondyle of the femur, movement arm along the fibula to lateral malleolus.
  Total eight treatment sessions will be given to each patient, and pre-treatment assessment will be done on very first day. Second assessment will be done on fourth treatment session, and final assessment will be on eighth treatment session.
Lower extremity functional scale (LEFS) | 6 weeks
  The Lower Extremity Functional Scale (LEFS) is a questionnaire containing 20 questions about a person's ability to perform everyday tasks. The LEFS can be used by clinicians as a measure of patients' initial function, ongoing progress and outcome, as well as to set functional goals. The resultant AKPS is a 13-item self-report questionnaire that evaluates subjective responses to specific activities and symptoms that are thought to correlate with anterior knee pain syndrome. The AKPS is scored from a minimum score of 0 to a maximum score of 100 points. This scale used for function of lower limb.
  Total eight treatment sessions will be given to each patient, and pre-treatment assessment will be done on very first day. Second assessment will be done on fourth treatment session, and final assessment will be on eighth treatment session.
Anterior knee pain scale (AKPS) | 6 weeks
  The resultant AKPS is a 13-item self-report questionnaire that evaluates subjective responses to specific activities and symptoms that are thought to correlate with anterior knee pain syndrome. The AKPS is scored from a minimum score of 0 to a maximum score of 100 points. This scale used for daily living performance status Total eight treatment sessions will be given to each patient, and pre-treatment assessment will be done on very first day. Second assessment will be done on fourth treatment session, and final assessment will be on eighth treatment session.

CONTACTS AND LOCATIONS:
Overall Officials: hassan javed, M.Phil(MSK), Principal Investigator — University of Lahore
Locations (1):
- PSRD hospital lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Petersen W, Ellermann A, Gosele-Koppenburg A, Best R, Rembitzki IV, Bruggemann GP, Liebau C. Patellofemoral pain syndrome. Knee Surg Sports Traumatol Arthrosc. 2014 Oct;22(10):2264-74. doi: 10.1007/s00167-013-2759-6. Epub 2013 Nov 13. PMID 24221245
- [Background] Yanez-Alvarez A, Bermudez-Pulgarin B, Hernandez-Sanchez S, Albornoz-Cabello M. Effects of exercise combined with whole body vibration in patients with patellofemoral pain syndrome: a randomised-controlled clinical trial. BMC Musculoskelet Disord. 2020 Aug 28;21(1):582. doi: 10.1186/s12891-020-03599-2. PMID 32859183
- [Background] Halabchi F, Abolhasani M, Mirshahi M, Alizadeh Z. Patellofemoral pain in athletes: clinical perspectives. Open Access J Sports Med. 2017 Oct 9;8:189-203. doi: 10.2147/OAJSM.S127359. eCollection 2017. PMID 29070955
- [Background] Smith BE, Selfe J, Thacker D, Hendrick P, Bateman M, Moffatt F, Rathleff MS, Smith TO, Logan P. Incidence and prevalence of patellofemoral pain: A systematic review and meta-analysis. PLoS One. 2018 Jan 11;13(1):e0190892. doi: 10.1371/journal.pone.0190892. eCollection 2018. PMID 29324820
- [Background] Lee JH, Jang KM, Kim E, Rhim HC, Kim HD. Effects of Static and Dynamic Stretching With Strengthening Exercises in Patients With Patellofemoral Pain Who Have Inflexible Hamstrings: A Randomized Controlled Trial. Sports Health. 2021 Jan/Feb;13(1):49-56. doi: 10.1177/1941738120932911. Epub 2020 Aug 13. PMID 32790575
- [Background] Xu X, Yao C, Wu R, Yan W, Yao Y, Song K, Jiang Q, Shi D. Prevalence of patellofemoral pain and knee pain in the general population of Chinese young adults: a community-based questionnaire survey. BMC Musculoskelet Disord. 2018 May 24;19(1):165. doi: 10.1186/s12891-018-2083-x. PMID 29793456
- [Background] Lankhorst NE, Bierma-Zeinstra SM, van Middelkoop M. Factors associated with patellofemoral pain syndrome: a systematic review. Br J Sports Med. 2013 Mar;47(4):193-206. doi: 10.1136/bjsports-2011-090369. Epub 2012 Jul 19. PMID 22815424
- [Background] Eng JJ, Pierrynowski MR. Evaluation of soft foot orthotics in the treatment of patellofemoral pain syndrome. Phys Ther. 1993 Feb;73(2):62-8; discussion 68-70. doi: 10.1093/ptj/73.2.62. PMID 8421719
- [Background] LaBella C. Patellofemoral pain syndrome: evaluation and treatment. Prim Care. 2004 Dec;31(4):977-1003. doi: 10.1016/j.pop.2004.07.006. PMID 15544830
- [Background] Powers CM, Landel R, Sosnick T, Kirby J, Mengel K, Cheney A, Perry J. The effects of patellar taping on stride characteristics and joint motion in subjects with patellofemoral pain. J Orthop Sports Phys Ther. 1997 Dec;26(6):286-91. doi: 10.2519/jospt.1997.26.6.286. PMID 9402564
- [Background] Tyler TF, Nicholas SJ, Mullaney MJ, McHugh MP. The role of hip muscle function in the treatment of patellofemoral pain syndrome. Am J Sports Med. 2006 Apr;34(4):630-6. doi: 10.1177/0363546505281808. Epub 2005 Dec 19. PMID 16365375
- [Background] Motealleh A, Kordi Yoosefinejad A, Ghoddosi M, Azhdari N, Pirouzi S. Trunk postural control during unstable sitting differs between patients with patellofemoral pain syndrome and healthy people: A cross-sectional study. Knee. 2019 Jan;26(1):26-32. doi: 10.1016/j.knee.2018.10.002. Epub 2018 Nov 22. PMID 30472048
- [Background] Khayambashi K, Mohammadkhani Z, Ghaznavi K, Lyle MA, Powers CM. The effects of isolated hip abductor and external rotator muscle strengthening on pain, health status, and hip strength in females with patellofemoral pain: a randomized controlled trial. J Orthop Sports Phys Ther. 2012 Jan;42(1):22-9. doi: 10.2519/jospt.2012.3704. Epub 2011 Oct 25. PMID 22027216
- [Background] Bolgla LA, Malone TR, Umberger BR, Uhl TL. Hip strength and hip and knee kinematics during stair descent in females with and without patellofemoral pain syndrome. J Orthop Sports Phys Ther. 2008 Jan;38(1):12-8. doi: 10.2519/jospt.2008.2462. Epub 2007 Nov 21. PMID 18349475
- [Background] Ireland ML, Willson JD, Ballantyne BT, Davis IM. Hip strength in females with and without patellofemoral pain. J Orthop Sports Phys Ther. 2003 Nov;33(11):671-6. doi: 10.2519/jospt.2003.33.11.671. PMID 14669962
- [Background] Callaghan MJ, Selfe J, McHenry A, Oldham JA. Effects of patellar taping on knee joint proprioception in patients with patellofemoral pain syndrome. Man Ther. 2008 Jun;13(3):192-9. doi: 10.1016/j.math.2006.11.004. Epub 2007 Feb 12. PMID 17296323